CLINICAL TRIAL: NCT02216201
Title: Clinical Utility of SUDOSCAN in the Pediatric Population
Status: Withdrawn | Type: Observational
Why Stopped: Sponsor terminated study
Sponsor: Impeto Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: Impeto-015
Record Dates: First submitted 2014-08-07; First posted 2014-08-13 (Estimated); Last update posted 2014-11-11 (Estimated); Status verified 2014-11

CONDITIONS: Childhood Obesity; Prediabetes; Diabetes
MeSH Terms: conditions — Pediatric Obesity; Prediabetic State; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The main purpose of this study is to evaluate whether SUDOSCAN is a valid, accurate clinical device for the the determination of sweat gland function in the pediatric population.

Primary Objective: To measure sweat gland function in a pediatric population

Secondary Objective: To determine thresholds on the SUDOSCAN scale for abnormal sweat gland function in the pediatric population

ELIGIBILITY:
Inclusion Criteria:

* Males and females ages 8 to 17 years
* Able to give assent as well as parental consent

Exclusion Criteria:

* History of type 1 or type 2 diabetes
* Chronic autoimmune condition
* Taking chronic immunosuppressive or anti-inflammatory medications
* Unable to apply palms of the hands and soles of the feet on the sensor plates during a 3 minute Sudoscan test
* Presence of hepatitis B or C
* Presence of HIV
* Presence of known neurological disorder
* Pregnancy and/or breastfeeding
* Any open wound on the soles of the feet or palms of the hands
* Participation in an ongoing clinical investigational drug trial
* Other serious medical conditions that in the opinion of the investigator, would compromise the subject's participation in the study

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 100 subjects will be recruited by age group, with approximately 10 subjects representative of each age between 8 and 17. Both lean and obese subjects will be included from University of Southern California's Childhood Obesity Research Center (CORC).
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-12; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Identification of participants with abnormal SUDOSCAN electrochemical skin conductance scores | Baseline
  * Sweat gland function will be assessed within each age group
  * Correlation with parameters associated with pre-diabetes and diabetes

CONTACTS AND LOCATIONS:
Locations (1):
- University of Southern California's Childhood Obesity Research Center (CORC), Los Angeles, California, United States

REFERENCES:
- [Background] Muller G, Olschewski J, Stange T, Hjellset VT, Bornstein S, Schwarz PE. Non-invasive screening of diabetes risk by assessing abnormalities of sudomotor function. Exp Clin Endocrinol Diabetes. 2015 Jan;123(1):34-8. doi: 10.1055/s-0033-1357128. Epub 2014 May 5. PMID 24798863
- [Background] Muller G, Parfentyeva E, Olschewsky J, Bornstein SR, Schwarz PE. Assessment of small fiber neuropathy to predict future risk of type 2 diabetes. Prim Care Diabetes. 2013 Dec;7(4):269-73. doi: 10.1016/j.pcd.2013.08.001. Epub 2013 Sep 27. PMID 24076379
- [Background] Chen L, Chen X, Ding R, Shi Q Jr, Hu D. Evaluation of EZSCAN as a screening tool for impaired glucose metabolism. Diabetes Res Clin Pract. 2013 May;100(2):210-4. doi: 10.1016/j.diabres.2013.03.001. Epub 2013 Mar 22. PMID 23529065